CLINICAL TRIAL: NCT05773495
Title: Implementation of Teleophthalmology in Urban Health Systems Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-0019; Ophthalmology (Other: UW Madison); 1UG1EY032446 (NIH)
Record Dates: First submitted 2023-03-02; First posted 2023-03-17 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Retinopathy
Keywords: screening
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual Care Followed by I-SITE Intervention (Experimental)
  Interventions: Other: I-SITE Intervention; Other: Usual Care Teleophthalmology

INTERVENTIONS:
Other: I-SITE Intervention — I-SITE is a coaching facilitated implementation program that guides clinical personnel through tailored integration of teleophthalmology into primary care workflows.
Other: Usual Care Teleophthalmology — All sites will initially receive usual care teleophthalmology, consisting of having an active teleophthalmology program located in the primary care clinic and access to the I-SITE online toolkit. All sites will utilize non-mydriatic retinal cameras (e.g. Topcon NW400) located in their primary care clinic to obtain a single 45-degree photo of the disc and macula with an anterior photo in each eye to provide diabetic eye screening as part of patients' usual care. Images are captured by trained primary care personnel and securely transmitted to eye doctors for evaluation.

SUMMARY:
This study is being conducted to test the effectiveness of I-SITE (Implementation for Sustained Impact in Teleophthalmology), an implementation program to sustain increased diabetic eye screening rates using teleophthalmology in urban, multi-payer health systems.

DETAILED DESCRIPTION:
The goal is to adapt I-SITE to a new population by identifying and testing strategies to overcome key barriers to teleophthalmology use among Latinos and Black Americans with diabetes.

The investigators will develop and test a culturally-adapted I-SITE intervention in urban, federally-qualified health centers serving low-income, Black and Latinx communities. The primary hypothesis is that the intervention will significantly increase the diabetic eye screening rate (primary outcome) at Access CHC and Outreach CHC at 6- and 12-months post-implementation compared to baseline. Secondary outcomes include monthly teleophthalmology use and follow-up rates for in-person eye care among screen positives. These data will facilitate rapid dissemination by helping key decision makers, such as health system administrators, determine whether to adopt the culturally-adapted I-SITE intervention.

The investigators are using a pre-post study design at each health system (site) to compare: (1) usual care teleophthalmology vs. the (2) I-SITE intervention.

1. Usual Care Teleophthalmology: All sites will initially receive usual care teleophthalmology, consisting of having an active teleophthalmology program located in the primary care clinic and access to the I-SITE online toolkit. The I-SITE online toolkit has been freely-available since December 2019 to all U.S. health systems and the general public. Health systems may also contact the study team for assistance with technical issues. All sites will utilize non-mydriatic retinal cameras (e.g. Topcon NW400) located in their primary care clinic to obtain a single 45-degree photo of the disc and macula with an anterior photo in each eye to provide diabetic eye screening as part of patients' usual care. Images are captured by trained primary care personnel and securely transmitted to eye doctors for evaluation. This workflow is based on existing protocols and guidelines set by the American Telemedicine Association Practice Recommendations for Diabetic Retinopathy.
2. I-SITE Intervention: Each site will subsequently receive all elements of usual care teleophthalmology plus the I-SITE implementation program. I-SITE is a coaching facilitated implementation program that guides clinical personnel through tailored integration of teleophthalmology into primary care workflows.

The I-SITE intervention includes:

* Initial 30-minute live webinar introduction and question & answer session between the I-SITE Coach and the participating primary care clinics.
* Two in-person 1-hour meetings between the I-SITE Coach and the local clinic team to discuss the teleophthalmology workflow, review current teleophthalmology use, diabetic eye screening rates, follow-up rates for in-person eye care among screen positives, set goals, and select implementation strategies to test. The meetings are to occur within 6 weeks after the introductory webinar.
* A series of 10 monthly teleconferences (15-30 min.) following the in-person meetings where the I-SITE Coach and local clinic team test and refine implementation strategies by reviewing data and providing feedback.

Two I-SITE Coaches will be present at all meetings (i.e., lead and assistant coach) to ensure continuity in case the lead I-SITE Coach is unexpectedly unable to attend a meeting.

I-SITE Coaches will also perform a half-day, on-site visit to physically walkthrough the teleophthalmology workflow, as well as meet with clinic administrators and staff, on the date of the first in-person meeting.

Data Collection Procedures:

Patient data will be collected within the established electronic health record at each participating health system as part of routine patient care, de-identified, and exported for secondary data analysis by clinic personnel at each health system who already have full access to their patient data as part of their employment, and regularly gather and report this type of data to health insurers as part of their clinical role (e.g., clinical quality improvement and electronic health record/information technology staff ). Personnel from each participating health system will only have access to data from their own health system.

ELIGIBILITY:
Inclusion Criteria:

* Eligible medical records will be identified using ICD-10 codes for diabetes type 1 or type 2
* Billing data will be identified using teleophthalmology (CPT codes 92228 or 92250)
* Identification of eligible records will be performed by clinic personnel at each health system who already have full access to their patient data as part of their employment, and regularly gather and report this type of data to health insurers as part of their clinical role

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in Diabetic Screening Rate | baseline (data is retrospective to evaluate pre-intervention beginning November 2022), 6 months post-intervention (up to 18 months), 12 months post-intervention (up to 24 months)
  Proportion of patients with diabetes with medical record documentation of diabetic eye screening within the last 12 months among patients with type 1 or type 2 diabetes who had at least 2 clinic visits with primary care provider within the past 24 months.

SECONDARY OUTCOMES:
Monthly Teleophthalmology Use | data collected monthly (retrospectively beginning November 2022 and up to 36 months prospectively)
  Monthly number of patients for whom an eye photo was ordered and for whom an eye photo was completed
Follow Up Rate For In-Person Eye Care Among Screen Positives | baseline (data is retrospective to evaluate pre-intervention beginning November 2022) and 12, 24, and 36 months
  Comparison of follow-up rates for in-person eye care among patients who have screened positive for ocular pathology requiring further in-person eye care on their teleophthalmology photos and subsequently obtained an in-person dilated eye exam with an eye care provider within 1 year of their teleophthalmology visit based on medical records review.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Liu, MD, MS, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data regarding patient demographics, whether they obtained diabetic eye screening, had teleophthalmology performed, any vision-threatening eye condition identified by teleophthalmology, and whether they followed-up for in-person eye care if they screened positive will be available to share.
Time Frame: up to 7 years after the completion of the primary outcome
Access Criteria: contact study PI for access

REFERENCES:
- See also: A Guide to Implementation for Sustained Impact in Teleophthalmology (I-SITE) — https://www.hipxchange.org/I-SITE